CLINICAL TRIAL: NCT00006152
Title: A Phase II, Restrictively Randomized, Open-Label, Pilot Study of Treatment Intensification of Early Virologic Failure
Brief Title: A Study to See If Taking One or Two Extra Drugs Can Lower HIV Levels in Patients Who Have Failed Their Anti-HIV Drug Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5061; 10898 (Registry Identifier: DAIDS ES); ACTG A5061; AACTG A5061
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; abacavir; amprenavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir

SUMMARY:
The purpose of this study is to see if adding 1 or 2 drugs to the anti-HIV therapy of patients whose HIV levels increased while taking their anti-HIV drugs can lower viral load (amount of HIV in the blood) and keep it low up to Week 24. (This study has been changed. Previously, only patients whose levels increased on their first round of anti-HIV drugs were being studied.) Anti-HIV drug treatments that contain a combination of 3 or more drugs can lower HIV levels, raise CD4 cell counts, and improve survival. Unfortunately, many patients "fail" their anti-HIV drug treatment when their HIV levels go above 500 copies/ml. Usually the next step is to switch the patient to different anti-HIV drugs. Doctors would like to see whether adding 1 or 2 different drugs to the "failed" treatment also can lower HIV levels. Adding 1 or 2 drugs might be better than switching all of the drugs since patients who take many different drugs can develop drug-resistant HIV. (This study has been changed. Previously, only patients taking protease inhibitors (PI) whose levels increased on their first round of anti-HIV drugs were being studied.)

DETAILED DESCRIPTION:
Successful therapy following viral rebound has been problematic. Intensification of the existing regimen by adding 1 or 2 drugs generally has been avoided. However, successfully adding new drugs to an existing regimen would be advantageous since it would expose the patient to fewer antiretroviral agents in the overall treatment course. Recent evidence suggests that a significant proportion of patients who experience viral rebound while receiving a protease inhibitor (PI) actually have viral rebound with a PI-sensitive virus. Other studies have shown that treatment decisions based on resistance assays result in better virologic outcomes. This trial examines further the effect of resistance assay-directed intensification of a PI-containing antiretroviral regimen on viral load. [AS PER AMENDMENT 04/03/01: The antiretroviral regimen need not contain a protease inhibitor.]

Patients are stratified by baseline plasma HIV-1 RNA levels (5,000 copies/ml or less versus greater than 5,000 copies/ml). Patients undergo phenotypic drug resistance testing prior to study entry. Based on the phenotypic results, patients are [AS PER AMENDMENT 11/9/00: selectively] randomized equally to 1 of 3 [AS PER AMENDMENT 11/9/00: 1 of 2] intensification strategies while remaining on their current, initial [AS PER AMENDMENT 11/9/00: (background)] antiretroviral therapy (ART). [AS PER AMENDMENT 04/03/01: ART need not be initial.] A patient is excluded from randomization to an arm if that arm contains a drug to which the patient has phenotypic resistance. Arm A adds abacavir (ABC). Arm B adds amprenavir (APV) [AS PER AMENDMENT 11/9/00: and ritonavir (RTV)]. Arm C adds didanosine (ddI) plus hydroxyurea (HU). [AS PER AMENDMENT 11/9/00: Arm C has been discontinued.] A patient's HIV must be sensitive to at least 3 drugs. [AS PER AMENDMENT 11/9/00: Each patient must be taking at least 3 drugs to which his/her HIV isolate is sensitive, including ABC or APV and at least 2 other drugs that are part of the current, initial (background) ART. If phenotypic resistance testing at screening indicates resistance to a nucleoside reverse transcriptase inhibitor (NRTI) drug in the patient's current, initial (background) ART, then the local investigator may choose to discontinue that drug. However, the patient and local investigator may choose to continue the drug but it will not be considered an active drug per this protocol.] [AS PER AMENDMENT 04/03/01: ART need not be initial.] Patients have regular clinic visits for physical exams and blood tests, including CD4 and CD8 cell counts, plasma HIV-1 RNA assays, and tests for pharmacokinetic variability. In the event of viral rebound of 500 copies/ml or more at Week 12 or later, phenotypic/genotypic drug resistance is assayed. In addition, phenotypic drug resistance is assayed at the primary endpoint (Week 24) and at the end of treatment (Week 48) on all patients.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are taking 3 or more anti-HIV drugs for at least 24 weeks. (This study has been changed. Previously, only patients taking their first round of anti-HIV drugs, which included a PI, were being studied.)
* Had a viral load below 500 copies/ml while on their anti-HIV drugs, and then had an increase in viral load to between 500 and 10,000 copies/ml. (This study has been changed. Previously, only patients whose levels increased on their first round of anti-HIV drugs were being studied.)
* Have a CD4 cell count of 100 cells/mm3 or more.
* Are age 13 or older (consent of a parent or legal guardian is required if under 18).
* Agree to use 2 methods of birth control during the study and for 60 days after. (This study has changed the birth control requirements.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are currently being treated for a serious infection or other serious medical illness.
* Have had certain illnesses in the past.
* Have a fever within 7 days of study entry.
* Have already taken all of the study drugs for more than 4 weeks.
* Are unable to take any of the study drugs.
* Have certain types of cancer.
* Received certain vaccines within 21 days of study entry.
* Have received certain medications.
* Are pregnant or breast-feeding.
* Patients will not be eligible for Group A if they:
* Have a history of hypersensitivity reaction to abacavir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, Study Chair; William Powderly, Study Chair; Mary Albrecht, Study Chair
Locations (13):
- United States (13):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Northwestern Univ Med School, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Beth Israel Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas